CLINICAL TRIAL: NCT04559282
Title: A Pivotal, Prospective, Single-centre, Randomized Test Order, Crossover, Open Label Study Comparing the Performance of a New Sound Processor With Unaided Hearing and Baha 5 in Adult Subjects With Conductive or Mixed Hearing Loss
Brief Title: Home Test of New Sound Processor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: Statistiska Konsultgruppen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CBAS5779
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Results first posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2020-12

CONDITIONS: Hearing Loss
Keywords: Conductive Hearing Loss; Mixed Hearing Loss
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New SP followed by Baha 5 SP followed by single blinded SP (Experimental): Aided hearing with new Sound Processor followed by aided hearing with the Baha 5 sound processor followed by unaided hearing followed by aided hearing with the new Sound Processor and Baha 5 in a laboratory environment (subject blinded for hearing testing).
  Interventions: Device: New Sound Processor
- Baha 5 SP followed by the New SP followed by single blinded SP (Experimental): Aided hearing with Baha 5 sound processor followed by aided hearing with the new Sound Processor followed by unaided hearing followed by aided hearing with the new Sound Processor and Baha 5 in a laboratory environment (subject blinded for hearing testing).
  Interventions: Device: New Sound Processor

INTERVENTIONS:
Device: New Sound Processor — The new Sound Processor is intended to be used as part of the Cochlear Baha System which uses bone conduction to transmit sounds to the cochlea. The New Sound Processor is indicated for patients with up to 55 dB sensorineural hearing loss.

SUMMARY:
The purpose of this clinical investigation is to test a new Sound Processor (SP) to compare hearing performance of the new Sound Processor with unaided hearing and Baha 5 SP in adult subjects and to investigate which device (new Sound Processor versus Baha 5) the subjects prefer.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject (18-<70 years of age)
* At least 12 months experience from using a Baha Connect system (percutaneous Baha)
* Subject with a conductive or mild to moderate mixed hearing loss. that would benefit from improved hearing from bone conduction device as judged by the research audiologist
* Willing and able to provide written informed consent

Exclusion Criteria:

* Signs of infection around the implant site
* Unable to follow investigational procedures
* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator
* Investigator site personnel directly affiliated with this investigation and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
* Cochlear employees
* Currently participating, or participated within the last 30 days, in another interventional clinical investigation/trial involving an investigational drug or device.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Ganlöv, MD, Study Director — Cochlear
Locations (1):
- Cochlear Bone Anchored Solutions AB (CBAS), Mölnlycke, Sweden

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for public sharing of IPD collected in this study. Data may be provided to individual researchers on request.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 participants were recruited in one centre from 23 September 2020 to 27 November 2020.
Groups:
- Baha 6 Max Followed by Baha 5 SP Followed by Unaided Hearing: Participants received Baha 6 Max followed by Baha 5 SP followed by Unaided
- Baha 5 SP Followed by Baha 6 Max Followed by Unaided Hearing: Participants received Baha 5 SP followed by Baha 6 Max followed by Unaided
Period: Intervention 1 (Day 0)
Arm/Group | Baha 6 Max Followed by Baha 5 SP Followed by Unaided Hearing | Baha 5 SP Followed by Baha 6 Max Followed by Unaided Hearing
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Intervention 2 (Day 7)
Arm/Group | Baha 6 Max Followed by Baha 5 SP Followed by Unaided Hearing | Baha 5 SP Followed by Baha 6 Max Followed by Unaided Hearing
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Intervention 3 (Day 14)
Arm/Group | Baha 6 Max Followed by Baha 5 SP Followed by Unaided Hearing | Baha 5 SP Followed by Baha 6 Max Followed by Unaided Hearing
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Crossover, participants received Baha 6 Max or Baha 5 SP followed by Baha 5 SP or Baha 6 Max followed by Unaided
Arm/Group | Entire Study Population
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 16

OUTCOME MEASURES:

1. Primary Outcome: Hearing Performance of Speech in Noise for Unaided Hearing and the Baha 6 Max Assessed Via Adaptive Speech Test in Noise
Description: Using validated lists of phonetically balanced sentences. Noise is kept constant at 65 dB Sound Pressure Level (SPL) and the speech is adapted stepwise to establish the speech-to-noise ratio providing a 50% level of understanding
Time Frame: Day 0, day 7 and day 14
Population: Data for Baha 6 Max was collected on Day 0 and day 7 for all 16 participants. Data for unaided hearing was collected on day 14 for all 16 participants.
Measure: Mean (Standard Deviation); unit: db SNR (decibel Speech in Noise Ratio)
Groups:
- Baha 6 Max: Baha 6 Max SP
- Unaided: Unaided hearing
Arm/Group | Baha 6 Max | Unaided
Number analyzed (Participants) | 16 | 16
db SNR (decibel Speech in Noise Ratio) | -3.7 (2.75) | 4.8 (6.55)

2. Primary Outcome: Participant Preference for the Baha 6 Max or Baha 5 SP Assessed Via Questions in the eCRF
Time Frame: Day 14
Population: Participants received Baha 6 Max or Baha 5 SP at day 0 followed by Baha 5 SP or Baha 6 Max at day 7
Measure: Count of Participants; unit: Participants
Groups:
- Baha 5: Baha 5 SP
Arm/Group | Baha 6 Max | Baha 5
Number analyzed (Participants) | 16 | 16
Participants | 13 | 3

3. Secondary Outcome: Descriptive Hearing Performance for the Baha 6 Max and Baha 5 SP in a Home/Normal Hearing Environment Assessed Via a Diary
Description: Diary completed by the participant with following topics: daily use of the sound processor (hours), change of battery, switch to their own sound processor.
Time Frame: Day 7 and day 14
Population: 16 participants assessed Baha 6 Max or Baha 5 SP at day 7 followed by Baha 5 SP or Baha 6 Max at day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Baha 6 Max | Baha 5
Number analyzed (Participants) | 16 | 16
Participants
  Daily use 10-16 hours | 13 | 9
  Daily use 6-8 hours | 2 | 6
  Daily use > 16 hours | 1 | 1
  Change battery in device | 2 | 8
  No change battery in device | 14 | 8
  Change to their own SP | 4 | 3
  No change to their own SP | 12 | 13

4. Secondary Outcome: Hearing Performance for the Baha 6 Max and Baha 5 SP Assessed Via Adaptive Speech Test in Noise
Description: Using validated lists of phonetically balanced sentences. Noise is kept constant at 65 dB SPL and the speech is adapted stepwise to establish the speech-to-noise ratio providing a 50% level of understanding
Time Frame: Day 0 and day 7
Population: 16 participants assessed Baha 6 Max or Baha 5 SP at day 0 followed by Baha 5 SP or Baha 6 Max at day 7
Measure: Mean (Standard Deviation); unit: dB SNR
Arm/Group | Baha 6 Max | Baha 5
Number analyzed (Participants) | 16 | 16
dB SNR | -3.7 (2.75) | -2.8 (2.44)

5. Secondary Outcome: Hearing Performance for the Baha 6 Max and Baha 5 SP Assessed Via Thresholds Audiometry
Description: Sound-field [0.25, 0.5, 1.0, 2.0, 3.0, 4.0, 6.0, 8.0 9.0 and 10.0 kHz]
Time Frame: Day 0 and day 7
Population: 16 participants assessed Baha 6 Max or Baha 5 SP at day 0 followed by Baha 5 SP or Baha 6 Max at day 7
Measure: Mean (Standard Deviation); unit: db HL (decibel Hearing Level)
Groups:
- Baha 5: Baha SP
Arm/Group | Baha 6 Max | Baha 5
Number analyzed (Participants) | 16 | 16
db HL (decibel Hearing Level)
  250 Hz | 29.7 (7.2) | 34.1 (8.2)
  500 Hz | 20.9 (9.4) | 24.1 (10.8)
  1000 Hz | 20.3 (8.8) | 23.1 (10.5)
  2000 Hz | 23.4 (11.4) | 25.3 (12.7)
  3000 Hz | 29.1 (15.4) | 33.4 (15.7)
  4000 Hz | 35 (14.1) | 37.5 (16.2)
  6000 Hz | 36.9 (15.2) | 39.7 (17.4)
  8000 Hz | 35.3 (120.0) | 56.9 (22.0)
  9000 Hz | 36.3 (20.0) | 65.3 (12.6)
  10000 Hz | 50.6 (19.8) | 65.3 (8.5)

6. Secondary Outcome: Hearing Performance for the Baha 6 Max and Baha 5 SP Assessed Via Speech Test in Quiet
Description: Using monosyllabic words presented at 65 dB SPL with scores recorded as % correct words.
Time Frame: Day 0 and day 7
Population: 16 participants assessed Baha 6 Max or Baha 5 SP at day 0 followed by Baha 5 SP or Baha 6 Max at day 7
Measure: Mean (Standard Deviation); unit: Percentage of correct words
Arm/Group | Baha 6 Max | Baha 5
Number analyzed (Participants) | 16 | 16
Percentage of correct words | 88.4 (14.4) | 77.9 (25.1)

7. Secondary Outcome: Hearing Performance for the Baha 6 Max and Baha 5 SP Assessed Via Participant Rating
Description: Participant rating on a likert scale from 1-5 where 1 represents the most negative and 5 represents the most positive experience of loudness, sound quality, sound clarity, speech understanding, presence of artefacts after listening to sound clips.
Time Frame: Day 14
Population: No data for speech understanding on sound clip 2 and for sound clarity on sound clip 1.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Baha 6 Max | Baha 5
Number analyzed (Participants) | 16 | 16
Score on a scale
  Loudness- sound clip 1 | 3.0 (0.5) | 2.6 (0.5)
  Loudness- sound clip 2 | 2.8 (0.9) | 2.6 (0.6)
  Artefacts- sound clip 1 | 4.69 (0.8) | 4.63 (1.1)
  Artefacts- sound clip 2 | 4.69 (0.5) | 4.5 (1.0)
  Speech understanding- sound clip 1 | 4.38 (0.89) | 3.63 (1.1)
  Sound quality- sound clip 1 | 4.25 (0.9) | 3.31 (1.2)
  Sound quality- sound clip 2 | 4.31 (0.7) | 3.44 (1.2)
  Sound clarity-sound clip 2 | 4.31 (0.9) | 3.19 (1.0)

8. Secondary Outcome: Hearing Performance for Baha 6 Max and Baha 5 SP Assessed Via Participant Rating for Internal Noise
Description: Participant rating Yes or No for internal noise after listening to sound clips.
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Baha 6 Max | Baha 5
Number analyzed (Participants) | 16 | 16
Participants
  Sound clip 1-Yes | 1 | 0
  Sound clip 1-No | 15 | 16
  Sound clip 2-Yes | 0 | 0
  Sound clip 2-No | 16 | 16

9. Secondary Outcome: Hearing Performance for Baha 6 Max and Baha 5 SP Assessed Via Participant Rating for Listening Effort.
Description: Participant rating for listening effort assessed with the Borg scale. The Borg scale measures the level of effort it takes trying to hear what is said in a sound clip. The scale is from 0-10 where 0= no effort at all and 10=maximal effort.
Time Frame: Day 14
Population: Data are for sound clip 1. No data available for sound clip 2.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Baha 6 Max | Baha 5
Number analyzed (Participants) | 16 | 16
Score on a scale | 1.97 (1.9) | 3.02 (2.6)

10. Secondary Outcome: Hearing Performance for Baha 6 Max and Unaided Assessed Via Thresholds Audiometry
Description: Sound-field [0.25, 0.5, 1.0, 2.0, 3.0, 4.0, 6.0, 8.0, 9.0 and 10.0 kHz]
Time Frame: Day 0, day 7 and day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: db HL (decibel Hearing Level)
Arm/Group | Baha 6 Max | Unaided
Number analyzed (Participants) | 16 | 16
db HL (decibel Hearing Level)
  250 Hz | 29.7 (7.2) | 46.3 (13.6)
  500 Hz | 20.9 (9.4) | 49.7 (12.0)
  1000 Hz | 20.3 (8.8) | 54.4 (12.6)
  2000 Hz | 23.4 (11.4) | 50.6 (50.6)
  3000 Hz | 29.1 (15.4) | 55.3 (16.4)
  4000 Hz | 35.0 (14.1) | 64.1 (17.8)
  6000 Hz | 36.9 (15.2) | 65.0 (18.4)
  8000 Hz | 35.3 (20.0) | 65.6 (17.3)
  9000 Hz | 36.3 (21.2) | 70.0 (15.5)
  10000 Hz | 50.6 (19.8) | 72.2 (10.3)

11. Secondary Outcome: Hearing Performance for Baha 6 Max and Unaided Assessed Via Speech Test in Quiet
Description: Using monosyllabic words presented at 65 dB SPL with scores recorded as % correct words
Time Frame: Day 0, day 7 and day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of correct words
Arm/Group | Baha 6 Max | Unaided
Number analyzed (Participants) | 16 | 16
Percentage of correct words | 88.4 (14.4) | 11 (21.8)

ADVERSE EVENTS:
Time Frame: 14 days
Description: Participants received Baha 6 Max or Baha 5 SP followed by Baha 5 SP or Baha 6 Max followed by Unaided
Arm/Group | Baha 6 Max | Baha 5 | Unaided
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT04559282/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT04559282/SAP_001.pdf